CLINICAL TRIAL: NCT01161030
Title: Almond Ingestion at Meal-time Reduces Postprandial Glycemia and Chronic Ingestion Reduces Hemoglobin A1c in Individuals With Well-controlled Type 2 Diabetes
Brief Title: Almonds and Diabetes Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Carol Johnston, Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: almond1
Record Dates: First submitted 2010-07-09; First posted 2010-07-13 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- almonds (Experimental): 1-oz raw almonds: 173 kcal, 4.6 g carbohydrate, 14.6 g fat
  Interventions: Dietary Supplement: Almonds
- Control (Placebo Comparator): cheese stick
  Interventions: Dietary Supplement: Almonds

INTERVENTIONS:
Dietary Supplement: Almonds

SUMMARY:
This trial examined the impact of acute and chronic almond ingestion on indicators of glucose control (postprandial glycemia and hemoglobin A1c). Hypotheses:

1. Almonds will stimulate the secretion of GLP-1 in healthy adults and in adults with T2D The investigators were not able to demonstrate a relationship between GLP-1 secretion and almond consumption. Individuals with T2D were characterized with significantly greater GLP-1 secretion than the non-diabetic control subjects.
2. Acute ingestion of almonds will decrease the postprandial glycemia and insulinemic responses in healthy controls and in individuals with T2D The investigators data support the hypothesis: almond consumption by individuals with T2D did attenuate postprandial glycemia; however, almond consumption did not alter glycemia in non-diabetic control subjects
3. Chronic almond ingestion for 12 weeks will reduce fasting glucose (FG) and A1c concentrations in individuals with T2D The investigators data demonstrated modest beneficial effect of almond consumption on A1c in individuals with T2D. Almond consumption was also associated with modest weight loss as compared to the control treatment (low fat cheese sticks).

ELIGIBILITY:
Inclusion Criteria:

* 12 subjects with diagnosed T2D for at least 1 year and 12 healthy individuals without T2D will be recruited for the acute almond trial.
* 24 subjects with diagnosed T2D for at least 1 year will be recruited for the chronic almond trial.
* Subjects from the campus population and nearby communities will be recruited to participate in these trials.
* Men and women must be willing to comply with the experimental protocol including the restriction of nut consumption:

  * subjects recruited for the acute almond study must agree not to consume any nuts or nut butters for 1-week prior to and during the 2-week trial
  * participants in the chronic almond study must agree not to consume nuts or nut butters more than 2 times per week during the 12 week trial.
* Participants must have a body mass index (BMI) from 20 to 35 kg/m2 and are aged 30 to 70 years.
* Subjects with T2D may take oral hyperglycemic agents.

Exclusion Criteria:

* Insulin use
* History of a peanut allergy
* Chronic or unresolved disease
* Current smoking habit
* Pregnant or lactating
* Medication use that may impact incretin secretion. [Incretins are gastrointestinal hormones secreted at meal-time.]

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-08; Primary Completion 2009-06 (Actual); Study Completion 2009-11 (Actual)